CLINICAL TRIAL: NCT05986825
Title: Validation of the French Version of the Score on Quality of Life (HiSQOL) in Hidradenitis Suppurativa (QUALIVER)
Acronym: QUALIVER
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0225 (QUALIVER)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-08

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients with Verneuil disease
  Interventions: Other: Verneuil questionnaire Validation

INTERVENTIONS:
Other: Verneuil questionnaire Validation — Request patient to Complete the questionnaire for validation of the French version

SUMMARY:
Validation of the French Version of the Score on Quality of Life in Hidradenitis Suppurativa. The French HiSQOL will be completed by 60 patients with hidradenitis suppurativa a first time, and a second time 1 week later.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient with Verneuil disease
* Beneficiary of or affiliated to a social security insurance
* Participation agreement

Exclusion Criteria:

* Patients physically or mentally unable to complete questionnaires.
* Refusal to participate
* Patient under legal protection (guardianship, curatorship) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Verneuil disease
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Validation of the questionnaire | During the visit and 1 week later

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: All collected data that underlie results in a publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.